CLINICAL TRIAL: NCT07387120
Title: Sertraline Dose and the Risk of Serious Adverse Events in Older Adults With Low Kidney Function: A Population-Based Cohort Study Research Protocol
Brief Title: Sertraline and the Risk of Serious Adverse Events
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 2025 0906 615 000_3; ICES # 2025 0906 615 000_3 (Other: ICES)
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease (CKD); Elderly; Outpatient
Keywords: Chronic Kidney Disease; High-throughput computing; Drug Adverse Events; Selective Serotonin Reuptake Inhibitors; Sertraline; Elderly; Geriatrics; Drug Safety
MeSH Terms: conditions — Renal Insufficiency, Chronic; Drug-Related Side Effects and Adverse Reactions | interventions — Sertraline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low dose of Sertraline (25 mg/day): Residents of Ontario (and possibly Alberta), aged 66 years or older with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for Sertraline (low-dose 25 mg/day) at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 01, 2008, to January 1, 2025, with a day supply of ≥7 days. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, and each patient will enter the cohort only once.
  Interventions: Drug: Sertraline 25 mg
- High dose of Sertraline (50 mg/day): Residents of Ontario (and possibly Alberta), aged 66 years or older with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for Sertraline (high-dose: 50 mg/day) at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 01, 2008, to January 1, 2025, with a day supply of ≥7 days. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, and each patient will enter the cohort only once.
  Interventions: Drug: Sertraline 50 mg

INTERVENTIONS:
Drug: Sertraline 50 mg — The primary exposure of interest will be oral Sertraline at a dose of 50 mg/day.
  Groups: High dose of Sertraline (50 mg/day)
Drug: Sertraline 25 mg — The primary exposure of interest will be oral Sertraline at a dose of 25 mg/day.
  Groups: Low dose of Sertraline (25 mg/day)

SUMMARY:
The goal of this population-based cohort study is to assess the safety of initiating a new outpatient prescription of 50 mg/day of Sertraline, a higher dose, compared to 25 mg/day, a lower dose, in adults aged 65+ with low kidney function. The primary question is whether initiating a new outpatient prescription of a higher dose of Sertraline (50mg/day) compared to a lower dose (25 mg/day) in older adults with low kidney function (an eGFR <45 mL/min per 1.73 m2, but not receiving dialysis or having a history of kidney transplantation) is associated with a higher 30-day risk. The outcome measured will be a composite of all-cause hospitalization, all-cause emergency department visit, or all-cause mortality.

DETAILED DESCRIPTION:
Background: Many older adults experience mental health disorders, such as depression and anxiety, alongside having low kidney function. Sertraline is a selective serotonin reuptake inhibitor. It is commonly prescribed to older adults for depression and anxiety treatment. However, aging and low kidney function can lead to increased plasma levels and a higher risk of adverse events. In prescribing references, product monographs, and other standard sources, inconsistent starting dose adjustments for patients with low kidney function have been noted. This inconsistency may contribute to the variable dosing observed in routine practice. Many older adults with low kidney function are initiated on sertraline at a dose of 50 mg per day. Compared to the lower dose of 25 mg per day, the higher dose may be associated with a higher rate of falls, fractures, gastrointestinal bleeding, arrhythmias, hospitalization, and mortality. Despite these concerns, there is a lack of real-world evaluation. The investigators used a novel high-throughput approach with Ontario healthcare databases. They identified an increased risk of adverse outcomes in patients with advanced CKD (estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m² without a history of dialysis or a kidney transplant) who were newly prescribed sertraline compared to a similar cohort of non-users. To build upon and validate these early findings, the investigators plan to conduct a population-based retrospective cohort study among older adults in Ontario, Canada. The study will use data to investigate the 30-day risk of serious adverse events after starting high versus low doses of sertraline in older adults with low kidney function. The aim is to enhance safer prescribing practices.

Methods: This population-based retrospective cohort study will include older adults (aged 66 years or older) with an estimated glomerular filtration rate (eGFR) less than 45 mL/min/1.73 m2, who are not receiving dialysis and have no history of kidney transplantation. Eligible participants will be identified from Ontario, and potentially Alberta, if they have been dispensed a new outpatient prescription for oral sertraline (25 or 50 mg/day) with a supply of at least seven days. In Ontario, participant accrual will occur from January 1, 2008, to January 1, 2025. Participants will be categorized into two groups based on the prescribed daily dose: low-dose (25 mg/day) and high-dose (50 mg/day). Propensity score weighting will be applied to achieve balance between groups across a comprehensive set of measured baseline characteristics. The primary outcome will be a 30-day composite of all-cause hospitalization, emergency department visit, or mortality.

Objectives: The study will assess whether initiation of a high dose (50 mg/day) compared to a low dose (25 mg/day) of sertraline is associated with a higher 30-day risk of a composite outcome (all-cause hospitalization, emergency department visit, or mortality) among older adults with low kidney function (eGFR <45 mL/min/1.73 m2, not on dialysis, no history of transplantation) in the outpatient setting. Additionally, the study will evaluate whether baseline eGFR category modifies the risk of the 30-day composite outcome among patients initiating higher versus lower doses of sertraline as outpatients. The cohort will be expanded to include all baseline eGFR levels, categorized as ≥60, 45-59, and <45 mL/min/1.73 m2.

Study Design and Setting: Data Sources: This study will employ a population-based retrospective cohort design using linked administrative health data from Ontario, Canada. If the Ontario cohort is insufficient to generate reliable estimates, the sample size will be augmented by conducting the same analysis using Alberta health administrative data. Ontario data will be obtained from ICES (ices.on.ca), which provides secure, encrypted individual-level data for Ontario residents, all of whom have universal access to hospital and physician services under a government-funded, single-payer healthcare system. Data use in this study is authorized under section 45 of Ontario's Personal Health Information Protection Act, which does not require review by a research ethics board. The study will utilize Ontario's comprehensive health databases, including the Ontario Drug Benefit (ODB) for prescription data, the Registered Persons Database (RPDB) for demographics and vital status, the Canadian Institute for Health Information Discharge Abstract Database (CIHI-DAD) and National Ambulatory Care Reporting System (NACRS) for hospitalizations and emergency visits, the Ontario Health Insurance Plan (OHIP) Database for physician billing claims, and the Ontario Laboratories Information System (OLIS) for laboratory data, including serum creatinine, to estimate kidney function. If the study is conducted in Alberta, data will be accessed through the Alberta Kidney Disease Network (AKDN), with the dataset available through approximately 2021. The study protocol, including the study description, design, and statistical analysis plan, will be publicly registered prior to conducting outcome analyses. Study results will be reported in accordance with RECORD reporting guidelines.

Study Population: The study will include all adults aged 66 years or older with an estimated glomerular filtration rate (eGFR) less than 45 mL/min per 1.73 m2. Individuals receiving dialysis or with a history of kidney transplantation will be excluded. Eligible participants must have received a new outpatient prescription for oral sertraline at an initial dose of 25 or 50 mg per day, with a supply of at least 7 days, between 2008 and 2024. The dispensing date of the prescription will define the index date. To ensure unique cohort entry, only the first eligible prescription per individual will be considered, and each person will be included in the cohort only once. Patients will be categorized as either high-dose or low-dose sertraline users.

Baseline Characteristics: Baseline variables will be obtained from health records, census files, hospital records, laboratory data, and physician claims. These variables will include demographic characteristics such as age, sex, rurality, and neighborhood income quintile, as well as comorbidities and medication use. Comorbidities and healthcare utilization will be assessed using 5-year and 1-year look-back periods from the index date, respectively. Medication use at baseline will be evaluated within 120 days prior to the index date. All participants must have an outpatient serum creatinine measurement within 365 days before cohort entry to enable estimation of eGFR using the 2021 CKD-EPI equation. Individuals with end-stage kidney disease, defined as those on dialysis or with a history of kidney transplantation, will be excluded.

Outcomes: The prespecified primary outcome is a 30-day composite outcome of all-cause hospitalization, emergency department visit, or mortality. Only the first hospitalization or emergency department visit within the initial 30 days is included. Each component of the primary composite outcome (all-cause hospitalization, all-cause emergency department visits, or all-cause mortality) is precisely coded in ICES data. The observation window for study outcomes commences on the date of prescription fill and extends for 30 days post-initiation. Loss to follow-up is anticipated to be less than 0.3% due to the observation window being under 90 days. In this age group, provincial emigration, which is the primary cause of loss to follow-up, occurs at a rate of less than 0.5% annually. Participant observation time will be censored at the earliest occurrence of the outcome of interest, death (if not the outcome of interest), or 30 days after the index date.

Secondary outcomes will include: (1) the individual components of the primary composite outcome (30-day all-cause hospitalization, all-cause emergency department visit, and all-cause mortality) analyzed separately; (2) a 30-day composite outcome of any hospital encounter (hospital admission or emergency department visit) involving delirium or encephalopathy, including disorientation, transient alteration of awareness, or other and unspecified symptoms affecting cognitive function, or a hospital encounter with receipt of an urgent computed tomography scan of the head; (3) a 30-day composite outcome of a hospital encounter (hospital admission or emergency department visit) with fracture (hip, femur, humerus, wrist/forearm, pelvis, and spine), falls, hypotension, or syncope; and (4) a 30-day hospital encounter (hospital admission or emergency department visit) with a composite outcome of atrial fibrillation/flutter, ventricular arrhythmia, or other arrhythmia, including pacemaker insertion, palpitations, unspecified tachycardia, atrioventricular block, supraventricular tachycardia, other conduction disorders, or implantable cardiac defibrillator.

Statistical analysis plan: Categorical variables will be summarized as frequencies and proportions. Continuous variables will be summarized as means with standard deviations (SD) or medians with interquartile ranges (IQR), as appropriate. Baseline characteristics will be compared between the high-dose (50 mg/day) and low-dose (25 mg/day) groups using standardized mean differences (SMDs). An absolute SMD greater than 10% will indicate a meaningful imbalance.

Balancing comparator group: Inverse probability of treatment weighting (IPTW) based on propensity scores will be used to balance baseline characteristics between the high-dose (50 mg/day) and low-dose (25 mg/day) groups, including known predictors of sertraline use. Propensity scores will be generated using a multivariable logistic regression model that includes all baseline characteristics. The average treatment effect in the treated (ATT) weights will be applied: patients in the low-dose group will receive weights calculated as (propensity score / [1 - propensity score]), and patients in the high-dose group will receive a weight of 1. This method will create a weighted pseudo-sample of low-dose sertraline (25 mg/day) patients with baseline characteristics similar to those in the high-dose sertraline (50 mg/day) group. Baseline characteristics will be compared between groups using standardized differences in both unweighted and weighted samples. Regression analysis: The primary composite outcome of all-cause hospitalization, all-cause emergency department visit, or all-cause mortality will be evaluated using modified Poisson regression to estimate the risk ratio (95% CI) and binomial regression to estimate the risk difference (95% CI) in the weighted cohort, with the low-dose sertraline (25 mg/day) group as the reference. Secondary analyses: All secondary outcomes will be tested independently without adjustment for multiple comparisons. Each test will be performed and reported separately. The primary outcome will be presented with its P-value, and all secondary outcomes will be reported as point estimates with 95% confidence intervals.

Additional analyses: The investigators will conduct five supplementary analyses. 1. Effect measure modification (EMM): The cohort will be expanded to include all estimated glomerular filtration rate (eGFR) levels, categorized into three groups: eGFR ≥60, 45-<60, and <45 mL/min/1.73 m². Baseline characteristics between high-dose (50 mg/day) and low-dose (25 mg/day) sertraline groups will be assessed using standardized differences, both for all renal function categories combined and within each eGFR category. To balance baseline characteristics between the high-dose and low-dose groups, the investigators will apply the inverse probability of treatment weighting (IPTW) method, based on propensity scores, for all eGFR categories combined and within each category. EMM will be evaluated on both additive and multiplicative scales. For additive interaction, binomial regression with an identity link will be used to estimate risk differences, including an interaction term between sertraline dose groups and eGFR strata. For multiplicative interaction, modified Poisson regression will estimate risk ratios, also including an interaction term between dose groups and eGFR strata. the estimated risk differences and risk ratio will be reported as point estimates with 95% confidence intervals. 2. A high-throughput computing analysis involving over 700 population-based, new-user cohort studies, each comparing 74 acute (30-day) outcomes across kidney function strata (PMID: 38186562), suggested that sertraline use versus non-use is associated with harm in patients with low kidney function. This analysis used Ontario data from January 1, 2008 to March 1, 2020. A subgroup analysis will be conducted for the primary analysis, restricting the cohort to periods before March 1, 2020 (overlapping with the high-throughput computing period) and after March 1, 2020 (no overlap). 3. Hazard ratios for all outcomes within 30 days will be computed to illustrate the effect of the intervention over time. Hazard ratios are expected to be similar to risk ratios. 4. E-value analyses will be performed to determine the minimum association strength an unmeasured confounder would require with both the prescription drug and the outcome to eliminate the observed association. 5. The risk of the primary outcome will be compared between new users of 50 mg/day sertraline and older adults with no sertraline use (non-users), as well as between new users of 25 mg/day sertraline and non-users. The same baseline characteristics and statistical analysis methods as in the primary analysis will be employed.

Combining Outcome Results from Ontario and Alberta. *This approach will be implemented only if analysis of Alberta data proceeds.* In Canada, individual-level patient data cannot be linked across provinces due to privacy regulations. To ensure data privacy and regulatory compliance, results from Ontario and Alberta will be combined using a privacy-preserving method. This method involves a single transfer of summary-level outputs from each province to the research team and will adapt techniques described by Shu et al. 2025.

ELIGIBILITY:
Inclusion Criteria:

Older adult aged 66 years or greater with low kidney function (an eGFR <45 mL/min per 1.73 m2 ) who have filled a new oral prescription for Sertraline at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program with a dose of 25 or 50 mg/day and a day supply of ≥7 days from January 1, 2008, to January 1, 2025 for Ontario (if needed, dates in Alberta to be finalized based on data availability). The investigators will exclude individuals undergoing dialysis or those who have received a kidney transplant. The age criterion is set to guarantee that individuals in this population had at least one year of prior universal outpatient prescription drug coverage. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, with each patient entering the cohort only once.

Exclusion Criteria:

1. Individuals with missing administrative database number, missing or invalid age (<0 or >105 years), missing or invalid sex, death on or before the index date, non-Ontario resident (for Ontario data).
2. Individuals less than 66 years of age on the index date.
3. Those with evidence of any study drug prescription 180 days before the index date (to restrict to new users only).
4. Individuals with other Selective Serotonin Reuptake Inhibitors (Citalopram, Escitalopram, Fluoxetine, Fluvoxamine, Paroxetine) prescription in the previous 180 days before the index date or on the index date.
5. Individuals with more than one study drug prescription on the index date, as this complicates the ability to ascertain the prescribed dose accurately.
6. Individuals with end-stage renal disease, chronic dialysis, or a kidney transplant prior to the index date.
7. Evidence with hospital discharge or emergency department visit in the two days prior to or on the index date to ensure a new outpatient prescription.
8. Individuals with no serum creatinine lab value in the 0-365 days prior to the index date.
9. Individuals with unstable baseline kidney function:

   * If the most recent serum creatinine test prior to the index date was an inpatient test [ER or hospitalization] (refer to this as test date 1), and there is not at least one 'outpatient' serum creatinine in the year before test date 1, OR
   * If the most recent prior serum creatinine test prior to the index date was an inpatient test [ER or hospitalization] (refer to this as test date 1), and while there is at least 'outpatient' serum creatinine test in the year before (test date 1), the most recent outpatient test prior to (test date 1) differs by an eGFR 10 mL/min/1.73 m2 or more from the value on (test date 1).

   In Ontario, it has been shown that an outpatient serum creatinine measurement in the province, conducted on a single occasion, usually represents a stable value.
10. Individuals receiving palliative care in the year prior to the index date, as in this setting dosing is less relevant; rather, the focus is comfort care. The investigators will restrict to the first prescription in individuals with more than one eligible prescription. Date of this prescription will be the index date (the date from which the outcomes start being assessed).

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults aged 66 years or older with low kidney function (eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new outpatient prescription for Sertraline with a dose of 25 or 50 mg/day and a day supply of ≥7 days between 2008 and 2024 in Ontario. The study accrual period for Alberta (if needed) will be determined based on data availability.
Sampling Method: Non-Probability Sample
Enrollment: 6893 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2025-01 (Actual); Study Completion 2026-01 (Actual)

PRIMARY OUTCOMES:
A composite outcome of all-cause hospitalization, all-cause emergency department visit, or all-cause mortality. | Older adults exposed to high-dose (50mg/day) vs low-dose (25 mg/day) Sertraline between Jan 1, 2008, and Jan 1,2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date
  All-cause hospitalization, all-cause emergency department visits, and all-cause mortality will be combined into a composite measure. Only the first hospitalization or first emergency department visit occurring after the cohort entry date will be considered.

SECONDARY OUTCOMES:
All-cause hospitalization | Exposed cohort to Sertraline (high dose (50mg/d) versus low dose (25 mg/d)) between January 1, 2008, and January 1, 2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date
  One of the components of the primary composite outcome, all-cause hospitalization, individually presented as a secondary outcome. Only the first hospitalization after the cohort entry date will be considered.
All-cause emergency department visit | Exposed cohort to Sertraline (high dose (50mg/d) versus low dose (25 mg/d)) between January 1, 2008, and January 1, 2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date
  One of the components of the primary composite outcome, all-cause emergency department visit, individually presented as a secondary outcome. Only the first emergency department visit after the cohort entry date will be considered.
All-cause mortality | Exposed cohort to Sertraline (high dose (50mg/d) versus low dose (25 mg/d)) between January 1, 2008, and January 1, 2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date
  One of the components of the primary composite outcome, all-cause mortality, individually presented as a secondary outcome.

OTHER OUTCOMES:
30-day hospital encounter with composite outcome of Atrial Fibrillation/flutter or ventricular arrhythmia or other arrhythmia | Exposed cohort to Sertraline (high dose (50mg/d) versus low dose (25 mg/d)) between January 1, 2008, and January 1, 2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  30-day hospital encounter (hospital admission or emergency visit) composite of atrial fibrillation/flutter or ventricular arrhythmia, or other arrhythmia (including pacemaker insertion, palpitations, tachycardia unspecified, atrioventricular block, supraventricular tachycardia, other conduction disorders, implantable cardiac defibrillator)
30-day composite outcome of a hospital encounter with delirium, encephalopathy, or hospital encounter with receipt of an urgent computed tomography scan of the head | Exposed cohort to Sertraline (high dose (50mg/d) versus low dose (25 mg/d)) between January 1, 2008, and January 1, 2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date
  30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with delirium or encephalopathy (disorientation, transient alteration of awareness, other and unspecified symptoms and signs involving cognitive function) or hospital admission with receipt of an urgent computed tomography scan of the head.
30-day composite outcome of a hospital encounter with fracture, falls, hypotension, or syncope | Exposed cohort to Sertraline (high dose (50mg/d) versus low dose (25 mg/d)) between January 1, 2008, and January 1, 2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date
  30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with fracture, falls, hypotension, or syncope.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Garg, Principal Investigator — London Health Sciences Centre Research Institute
Locations (1):
- London Health Sciences Centre Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The dataset in Ontario from this study is held securely in coded form at ICES. While legal data sharing agreements between ICES and data providers (e.g., healthcare organizations and government) prohibit ICES from making the dataset publicly available, access may be granted to those who meet pre-specified criteria for confidential access, available at www.ices.on.ca/DAS (email: das@ices.on.ca). The full dataset creation plan and underlying analytic code may be available from the authors all secondary outcomes will be reported as point estimates with 95% confidence intervals upon request, understanding that the computer programs may rely upon coding templates or macros that are unique to ICES and are therefore either inaccessible or may require modification.

REFERENCES:
- [Background] Abdullah SS, Rostamzadeh N, Muanda FT, McArthur E, Weir MA, Sontrop JM, Kim RB, Kamran S, Garg AX. High-Throughput Computing to Automate Population-Based Studies to Detect the 30-Day Risk of Adverse Outcomes After New Outpatient Medication Use in Older Adults with Chronic Kidney Disease: A Clinical Research Protocol. Can J Kidney Health Dis. 2024 Jan 6;11:20543581231221891. doi: 10.1177/20543581231221891. eCollection 2024. PMID 38186562